CLINICAL TRIAL: NCT01107925
Title: A Pharmacokinetic and Pharmacodynamic Comparison of Prasugrel and Clopidogrel in Low Body Weight Versus Higher Body Weight Aspirin-Treated Subjects With Stable Coronary Artery Disease
Brief Title: Comparison of Prasugrel and Clopidogrel in Low Body Weight Versus Higher Body Weight With Coronary Artery Disease
Acronym: FEATHER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12921; H7T-MC-TADI (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease
Keywords: Platelet function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mg prasugrel (Experimental)
  Interventions: Drug: prasugrel
- 10 mg prasugrel (Active Comparator)
  Interventions: Drug: prasugrel
- 75 mg clopidogrel (Active Comparator)
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: prasugrel — Administered orally, daily for 12 days
  Other Names: Efient; Effient; LY640315; CS747
  Arms: 10 mg prasugrel; 5 mg prasugrel
Drug: clopidogrel — Administered orally, daily for 12 days
  Arms: 75 mg clopidogrel

SUMMARY:
The 5-milligram (mg) dose of prasugrel in low body weight (LBW) patients with coronary artery disease produces a pharmacodynamic response within the same therapeutic range as 10-mg dose in higher body weight (HBW) patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of stable coronary artery disease who are not currently indicated for treatment with a thienopyridine (that is, prasugrel, clopidogrel, or ticlopidine)
* Provision of written informed consent
* For women of child-bearing potential only (that is, women who are not surgically or chemically sterilised and who are between menarche and 1 year post menopause), test negative for pregnancy (based on a urine or serum pregnancy test to be performed before randomisation) and agree to use a reliable method of birth control during the study

Exclusion Criteria:

* Unstable coronary artery disease
* Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Graft Surgery (CABG) within the previous 90 days
* History of refractory ventricular arrhythmias within the last 6 months; an implanted defibrillator device; congestive heart failure within 6 months prior to screening; major surgery, or severe trauma, fracture or organ biopsy within 3 months prior to enrollment
* Any planned surgical procedure or any coronary revascularisation (surgical or percutaneous) planned within 60 days following randomisation
* Any known contraindication to treatment with an antiplatelet agent
* Significant hypertension at the time of screening or randomisation
* Clinically significant out-of-range values for platelet count or haemoglobin at screening, in the investigator's opinion, or results of clinical laboratory tests at the time of screening that are judged to be clinically significant for the study population, as determined by the investigator
* Prior history or presence of significant bleeding disorders, abnormal bleeding tendency, or personal history of coagulation or bleeding disorders.
* Prior history or clinical suspicion of cerebral vascular malformations, intracranial neoplasm, Transient Ischemic Attack (TIA) or stroke.
* Prior history of thrombocytopenia or thrombocytosis
* Use of antiplatelet agents (besides aspirin) within 10 days prior to screening; the use (or planned use) of heparin, oral anticoagulants, or fibrinolytic agents within 30 days of screening; or subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDS) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dublin, Ireland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nieuwegein, Netherlands
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala

REFERENCES:
- [Derived] Jakubowski JA, Angiolillo DJ, Zhou C, Small DS, Moser BA, Ten Berg JM, Brown PB, James S, Winters KJ, Erlinge D. The influence of body size on the pharmacodynamic and pharmacokinetic response to clopidogrel and prasugrel: a retrospective analysis of the FEATHER study. Thromb Res. 2014 Sep;134(3):552-7. doi: 10.1016/j.thromres.2014.05.019. Epub 2014 May 21. PMID 25022828
- [Derived] Erlinge D, Ten Berg J, Foley D, Angiolillo DJ, Wagner H, Brown PB, Zhou C, Luo J, Jakubowski JA, Moser B, Small DS, Bergmeijer T, James S, Winters KJ. Reduction in platelet reactivity with prasugrel 5 mg in low-body-weight patients is noninferior to prasugrel 10 mg in higher-body-weight patients: results from the FEATHER trial. J Am Coll Cardiol. 2012 Nov 13;60(20):2032-40. doi: 10.1016/j.jacc.2012.08.964. Epub 2012 Oct 17. PMID 23083774

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mg Prasugrel (LBW): During Study Period 1, participants received the 5-milligram (mg) prasugrel dose for 12 days without intervening or terminal washout periods. Participants in the low body weight (LBW; <60 kilograms [kg]) treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2.
- 10 mg Prasugrel (LBW): Participants in the LBW treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
- 75 mg Clopidogrel (LBW): Participants in the LBW treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 75-mg clopidogrel or 10-mg prasugrel dose during Study Period 2 or Study Period 3.
- 5 mg Prasugrel (HBW): Participants in the higher body weight (HBW; ≥ 60 kg) treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 5-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
- 10 mg Prasugrel (HBW): During Study Period 1, participants in the HBW treatment sequence received the 10-mg prasugrel dose for 12 days without intervening or terminal washout periods.
- 75 mg Clopidogrel (HBW): Participants in the HBW treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
Period: Period 1-Randomization up Through Day 12
Arm/Group | 5 mg Prasugrel (LBW) | 10 mg Prasugrel (LBW) | 75 mg Clopidogrel (LBW) | 5 mg Prasugrel (HBW) | 10 mg Prasugrel (HBW) | 75 mg Clopidogrel (HBW)
Started | 34 | 0 | 0 | 0 | 38 | 0
Took at Least 1 Dose of Study Drug | 34 | 0 | 0 | 0 | 38 | 0
Completed | 33 | 0 | 0 | 0 | 37 | 0
Not Completed | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | 5 mg Prasugrel (LBW) | 10 mg Prasugrel (LBW) | 75 mg Clopidogrel (LBW) | 5 mg Prasugrel (HBW) | 10 mg Prasugrel (HBW) | 75 mg Clopidogrel (HBW)
Started | 0 (5 mg prasugrel (Period 1, LBW treatment) switched to 10 mg prasugrel or 75 mg clopidogrel (Period 2)) | 16 | 17 | 20 | 0 (10 mg prasugrel (Period 1, HBW treatment) switched to 5 mg prasugrel or 75 mg clopidogrel (Period 2)) | 17
Took at Least 1 Dose of Study Drug | 0 | 16 | 17 | 20 | 0 | 17
Completed | 0 | 15 | 17 | 20 | 0 | 16
Not Completed | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | 5 mg Prasugrel (LBW) | 10 mg Prasugrel (LBW) | 75 mg Clopidogrel (LBW) | 5 mg Prasugrel (HBW) | 10 mg Prasugrel (HBW) | 75 mg Clopidogrel (HBW)
Started | 0 | 17 (75 mg clopidogrel (Period 2, LBW treatment sequence) crossed over to 10 mg prasugrel (Period 3).) | 15 (10 mg prasugrel (Period 2, LBW treatment sequence) crossed over to 75 mg clopidogrel (Period 3).) | 16 (75 mg clopidogrel (Period 2, HBW treatment sequence) crossed over to 5 mg prasugrel (Period 3).) | 0 | 20 (5 mg prasugrel (Period 2, HBW treatment sequence) crossed over to 75 mg clopidogrel (Period 3).)
Took at Least 1 Dose of Study Drug | 0 | 17 | 15 | 16 | 0 | 20
Completed | 0 | 17 | 15 | 16 | 0 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Sequence: Pras 5mg, Pras 10mg, Clop 75mg (LBW): Participants in the low body weight (LBW; <60 kilograms [kg]) group received 5 milligrams (mg) of Prasugrel (Pras) during Study Period 1, followed by 10 mg Pras in Study Period 2, followed by 75 mg clopidogrel (Clop) in Study Period 3.
- Dose Sequence: Pras 5mg, Clop 75 mg, Pras 10mg (LBW): Participants in the LBW group received 5 mg Pras during Study Period 1, followed by 75 mg Clop in Study Period 2, and 10 mg Pras in Study Period 3.
- Dose Sequence: Pras 10mg, Pras 5mg, Clop 75 mg (HBW): Participants in the higher body weight (HBW; ≥60 kg) group received 10 mg Pras during Study Period 1, followed by 5 mg Pras in Study Period 2, followed by 75 mg Clop in Study Period 3.
- Dose Sequence: Pras 10mg, Clop 75 mg, Pras 5mg (HBW): Participants in the HBW group received 10 mg Pras during Study Period 1, followed by 5 mg Pras in Study Period 2, followed by 75 mg Clop in Study Period 3.
- Total: Total of all reporting groups
Arm/Group | Dose Sequence: Pras 5mg, Pras 10mg, Clop 75mg (LBW) | Dose Sequence: Pras 5mg, Clop 75 mg, Pras 10mg (LBW) | Dose Sequence: Pras 10mg, Pras 5mg, Clop 75 mg (HBW) | Dose Sequence: Pras 10mg, Clop 75 mg, Pras 5mg (HBW) | Total
Number analyzed (Participants) | 17 | 17 | 21 | 17 | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.07) | 63.2 (7.65) | 61.4 (9.57) | 64.6 (6.91) | 62.6 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 7 | 5 | 41
  Male | 2 | 3 | 14 | 12 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 8 | 11 | 8 | 37
  Unknown or Not Reported | 7 | 9 | 10 | 9 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 3 | 4
  White | 17 | 16 | 20 | 14 | 67
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 2 | 2 | 4
  Ireland | 2 | 2 | 8 | 6 | 18
  Netherlands | 9 | 8 | 5 | 5 | 27
  Sweden | 6 | 7 | 6 | 4 | 23
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 56.06 (4.575) | 56.78 (2.619) | 83.60 (17.146) | 85.96 (11.898) | 71.33 (17.980)
Tobacco Use Status [Number; unit: participants]
  Tobacco Use Yes | 7 | 8 | 5 | 4 | 24
  Tobacco Use No | 10 | 9 | 16 | 13 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximum Platelet Aggregation (MPA) to 20 Micromolar (µM) Adenosine Diphosphate (ADP) at Day 12 (Period 1)
Description: MPA to 20 micromolar (μM) ADP was assessed by light transmission aggregometry (LTA), an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance). A lower MPA reflects stronger platelet inhibition, whereas a higher MPA reflects weaker inhibition.
Time Frame: Baseline, Day 12
Population: Primary intent-to-treat (ITT) pharmacodynamic (PD) population: all randomized participants who continued in the study through Day 12, and had at least 1 evaluable PD assessment at Day 12. Participants were analyzed based on the treatment group they were randomized to irrespective to the treatment they received.
Measure: Median (Inter-Quartile Range); unit: percent aggregation
Groups:
- Prasugrel 5 mg (LBW): Participants in the low body weight (LBW; <60 kilograms [kg]) group received the 5-milligram (mg) prasugrel dose in Study Period 1.
- Prasugrel 10 mg (HBW): Participants in the higher body weight (HBW; ≥60 kg) group received the 10-mg prasugrel dose in Study Period 1.
Arm/Group | Prasugrel 5 mg (LBW) | Prasugrel 10 mg (HBW)
Number analyzed (Participants) | 33 | 37
percent aggregation
  Baseline | 75.00 [70.00 to 80.00] | 76.40 [71.00 to 84.10]
  Day 12 (n=32, 37) | 47.00 [37.70 to 56.45] | 47.00 [39.00 to 57.10]
Statistical Analysis 1: Comparison: Prasugrel 5 mg (LBW) vs Prasugrel 10 mg (HBW); Test type: Non-Inferiority or Equivalence — Difference in median MPA in response to 20 μM ADP in LBW participants who received 5 mg prasugrel to the 75th percentile of MPA response to 20 μM ADP in HBW participants who received10 mg prasugrel at the end of Study Period 1 (Baseline through Day 12) was estimated from the observed data; p = 0.526, bootstrap (to determine 95% CI); Estimate of the difference = -10.10, 95% CI 2-sided [-23.40 to 0.20] — Estimate of the difference = [median (low body weight) - Q3 (higher body weight)]

2. Secondary Outcome: Change From Baseline in Vasodilator-Associated Stimulated Phosphoprotein (VASP) at Day 12 of Therapy
Description: VASP phosphorylation levels, expressed as the platelet reactivity index (PRI), reflect the degree of thienopyridine-mediated P2Y12 receptor inhibition and were used to compare prasugrel versus clopidogrel, in low body weight (LBW) participants compared to higher body weight (HBW) participants. PRI was calculated by VASP. The PRI indicates the level of P2Y12 receptor inhibition. A lower PRI reflects stronger inhibition of P2Y12 receptor thus stronger platelet inhibition, whereas a higher PRI reflects weaker inhibition of P2Y12 receptor and weaker platelet inhibition.
Time Frame: Baseline, Day 12
Population: As-treated pharmacodynamic (PD) population: all randomized participants who received at least 1 dose of study drug and provided at least 1 evaluable PD measure at 1 of the 3 periods. Participants were analyzed based on the treatment they received for each period regardless of their randomized treatment assignment.
Measure: Mean (Standard Deviation); unit: percentage PRI
Groups:
- 75 mg Clopidogrel (HBW): Participants in the HBW treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 75-mg clopidogrel or 5-mg prasugrel dose either during Study Period 2 or Study Period 3.
Arm/Group | 5 mg Prasugrel (LBW) | 10 mg Prasugrel (LBW) | 75 mg Clopidogrel (LBW) | 5 mg Prasugrel (HBW) | 10 mg Prasugrel (HBW) | 75 mg Clopidogrel (HBW)
Number analyzed (Participants) | 33 | 32 | 32 | 36 | 37 | 36
percentage PRI
  Baseline | 86.57 (4.44) | 86.44 (4.45) | 86.44 (4.45) | 86.77 (3.42) | 86.76 (3.37) | 86.77 (3.42)
  Day 12 (n=32,31,30,32,36,34) | 33.54 (15.77) | 15.09 (11.71) | 39.01 (17.49) | 56.87 (15.47) | 27.79 (18.13) | 56.35 (18.33)

3. Secondary Outcome: Change From Baseline in VerifyNow® P2Y12 Reaction Units (PRU) at Day 12 of Therapy
Description: The Accumetrics VerifyNow® P2Y12 assay measures platelet aggregation in whole blood and is reported in PRU. PRU indicates the extent of P2Y12 receptor-mediated platelet aggregation calculated as a function of rate and extent of platelet aggregation in an adenosine phosphate (ADP)-containing channel of the device. A lower PRU reflects stronger inhibition of platelet aggregation, whereas a higher PRU reflects weaker inhibition of platelet aggregation.
Time Frame: Baseline, Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: P2Y12 reaction units (PRU)
Groups:
- 5 mg Prasugrel (LBW): During Study Period 1, participants received the 5-milligram (mg) prasugrel dose for 12 days without intervening or terminal washout periods. Participants in the low body weight (LBW; (<60 kilograms [kg]) treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2.
- 75 mg Clopidogrel (HBW): Participants in the HBW treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 75-mg clopidogrel or 5-mg prasugrel dose during Study Period 2 or Study Period 3.
Arm/Group | 5 mg Prasugrel (LBW) | 10 mg Prasugrel (LBW) | 75 mg Clopidogrel (LBW) | 5 mg Prasugrel (HBW) | 10 mg Prasugrel (HBW) | 75 mg Clopidogrel (HBW)
Number analyzed (Participants) | 33 | 32 | 32 | 36 | 37 | 36
P2Y12 reaction units (PRU)
  Baseline | 317.9 (46.10) | 315.3 (44.26) | 315.3 (44.26) | 312.8 (43.01) | 311.0 (43.76) | 312.8 (43.01)
  Day 12 (n=32,31,32,35,34,34) | 129.5 (62.14) | 55.9 (38.08) | 151.7 (57.46) | 193.9 (74.09) | 102.1 (69.49) | 207.0 (67.62)

4. Secondary Outcome: Pharmacokinetic (PK) Analysis of the Concentration-Time Curve (AUC)
Description: A pharmacokinetic-pharmacodynamic (PK-PD) analysis comparing MPA (LTA) and AUC was conducted as originally intended, however the graphic output is not possible here. Therefore, the PK portion is presented here as AUC and the PD portion is presented in Secondary Outcome Measure #5. AUC was calculated through the last scheduled sampling time of 4 hours [AUC (0-4)] or through the sampling time of the last quantifiable concentration prior to 4 hours. AUC values were denoted AUC(0-tlast) in both instances.
Time Frame: baseline (pre-dose) up to 4 hours post-dose
Population: All available PK sample data from all treated participants who contributed complete PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram•hour/milliliter (ng•hr/mL)
Units Other Than Participants: Participant Profiles
Groups:
- Prasugrel 5 mg (LBW): During Study Period 1, participants received the 5-milligram (mg) prasugrel dose for 12 days without intervening or terminal washout periods. Participants in the low body weight (LBW; <60 kilograms [kg]) treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2.
- Prasugrel 10 mg (LBW); Clopidogrel 75 mg (LBW): Participants in the LBW treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
- Prasugrel 5 mg (HBW): Participants in the higher body weight (HBW; ≥ 60 kg)treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 5-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
- Prasugrel 10 mg (HBW): During Study Period 1, participants in the HBW treatment sequence received the 10-mg prasugrel dose for 12 days without intervening or terminal washout periods.
- Clopidogrel 75 mg (HBW): Participants in the HBW treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
Arm/Group | Prasugrel 5 mg (LBW) | Prasugrel 10 mg (LBW) | Clopidogrel 75 mg (LBW) | Prasugrel 5 mg (HBW) | Prasugrel 10 mg (HBW) | Clopidogrel 75 mg (HBW)
Number analyzed (Participants) | 34 | 33 | 30 | 36 | 38 | 37
Number analyzed (Participant Profiles) | 34 | 50 | 45 | 52 | 38 | 57
nanogram•hour/milliliter (ng•hr/mL) | 28.9 (37) | 59.3 (40) | 18.4 (38) | 19.4 (46) | 46.7 (44) | 12.7 (60)

5. Secondary Outcome: Change From Baseline in Maximum Platelet Aggregation (MPA) as Measured by Light Transmission Aggregometry (LTA) at Day 12 of Therapy
Description: MPA to 20 micromolar (μM) adenosine diphosphate (ADP) was assessed by LTA, an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance). A lower MPA reflects stronger platelet inhibition, whereas a higher MPA reflects weaker inhibition.
Time Frame: Baseline , Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent aggregation
Groups:
- 75 mg Clopidogrel (LBW): Participants in the LBW treatment sequence in Period 1 (on 5 mg prasugrel) were switched to either the 10-mg prasugrel or the 75-mg clopidogrel dose for Period 2 or Period 3.
- 5 mg Prasugrel (HBW): Participants in the higher body weight (HBW; ≥ 60 kg)treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 5-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
- 10 mg Prasugrel (HBW): During Study Period 1, participants in the (HBW; ≥ 60 kg) treatment sequence received the 10-mg prasugrel dose for 12 days without intervening or terminal washout periods.
- 75 mg Clopidogrel (HBW): Participants in the HBW treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either 5-mg prasugrel or the 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
Arm/Group | 5 mg Prasugrel (LBW) | 10 mg Prasugrel (LBW) | 75 mg Clopidogrel (LBW) | 5 mg Prasugrel (HBW) | 10 mg Prasugrel (HBW) | 75 mg Clopidogrel (HBW)
Number analyzed (Participants) | 33 | 32 | 32 | 36 | 37 | 36
percent aggregation
  Baseline | 76.27 (9.49) | 76.20 (9.63) | 76.20 (9.63) | 77.63 (12.29) | 77.93 (12.27) | 77.63 (12.29)
  Day 12 ( n= 32,32,31,35,37,35) | 48.10 (13.89) | 38.11 (14.17) | 51.41 (13.56) | 61.90 (18.93) | 47.92 (15.18) | 65.28 (17.83)

ADVERSE EVENTS:
Groups:
- 5 mg Prasugrel (LBW): During Study Period 1, participants received 5 milligrams (mg) prasugrel for 12 days without intervening or terminal washout periods. Participants in the low body weight (LBW; <60 kilograms [kg]) treatment sequence in Study Period 1 (5 mg prasugrel) were switched to either the 10-mg prasugrel or 75-mg clopidogrel dose during Study Period 2.
- 5 mg Prasugrel (HBW): Participants in the higher body weight (HBW; ≥ 60 mg) treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 5-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
- 75 mg Clopidogrel (HBW): Participants in the HBW treatment sequence in Study Period 1 (10 mg prasugrel) were switched to either the 5-mg prasugrel or 75-mg clopidogrel dose during Study Period 2 or Study Period 3.
Arm/Group | 5 mg Prasugrel (LBW) | 10 mg Prasugrel (LBW) | 75 mg Clopidogrel (LBW) | 5 mg Prasugrel (HBW) | 10 mg Prasugrel (HBW) | 75 mg Clopidogrel (HBW)
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/33 | 0/32 | 0/36 | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 20/34 | 21/33 | 14/32 | 10/36 | 12/38 | 14/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Prasugrel (LBW) (N=34) | 10 mg Prasugrel (LBW) (N=33) | 75 mg Clopidogrel (LBW) (N=32) | 5 mg Prasugrel (HBW) (N=36) | 10 mg Prasugrel (HBW) (N=38) | 75 mg Clopidogrel (HBW) (N=37)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — This event occurred after study completion, but within the 30 day follow-up period. This was the last treatment assigned for this participant.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Prasugrel (LBW) (N=34) | 10 mg Prasugrel (LBW) (N=33) | 75 mg Clopidogrel (LBW) (N=32) | 5 mg Prasugrel (HBW) (N=36) | 10 mg Prasugrel (HBW) (N=38) | 75 mg Clopidogrel (HBW) (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 9 (9) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Formication (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 5 (7) | 3 (7) | 5 (7) | 3 (4) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days